CLINICAL TRIAL: NCT00248963
Title: A Multicenter, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Levonorgestrel 90 Mg and Ethinyl Estradiol 20 Mg in a Continuous 28-Day Regimen for Oral Contraception Versus a Cyclic 21-Day Regimen Oral Contraceptive
Brief Title: Study Evaluating Levonorgestrel and Ethinyl Estradiol in Oral Contraception
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 0858A2-315
Record Dates: First submitted 2005-11-02; First posted 2005-11-04 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2006-05

CONDITIONS: Oral Contraceptive
Keywords: Oral Contraceptive
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol

INTERVENTIONS:
Drug: Levonorgestrel 90 mg and Ethinyl Estradiol 20 mg

SUMMARY:
To evaluate the contraceptive efficacy of an oral contraceptive containing a combination of LNG 90 mg/EE 20 mg in a continuous-use regimen and to evaluate the safety compared to LNG 100 mg/EE 20 mg for 21 days followed by a 7-day hormone-free interval in a cyclic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18 to 49 years who are willing to rely upon a combination birth control pill as their only method of contraception.
* Women must be sexually active and at risk for becoming pregnant.
* Women must have had regular (21- to 35- day) menstrual cycles for the 3-month period preceding study visit 1.

Exclusion Criteria:

* High blood pressure
* Age greater then 34 and smoking more than 15 cigarettes per day.
* Depression requiring hospitalization or associated with suicidal ideation within the last 3 years.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600
Dates: Study Completion 2004-10

PRIMARY OUTCOMES:
To evaluate the contraceptive efficacy of an OC containing a combination of LNG 90 mg/EE 20 mg in a continuous-use regimen and the safety compared to LNG 100 mg/EE 20 mg for 21 days followed by a 7-day hormone-free interval in a cyclic regimen

SECONDARY OUTCOMES:
To evaluate the effects on vaginal bleeding profile, hemostatic balance, lipid, carbohydrate, bone metabolism measures, hemoglobin levels, discontinuation rates, compliance with respect to pill taking, subject satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer